CLINICAL TRIAL: NCT05746286
Title: Continuous, Real-time, Remote Monitoring of Vital Signs With Telehealth to Prevent Readmissions for Dysglycemia: Discharge Remote Monitoring System (DIREMOS)
Brief Title: Remote Monitoring of Vital Signs With Telehealth to Prevent Readmissions for Dysglycemia
Acronym: DIREMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL-1000045
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Dysglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Criteria Met (Other): Participants will be provided continuous vitals and glucose monitors at hospital discharge for their treating physician to have access to the data to review
  Interventions: Device: Dexcom G6 CGM

INTERVENTIONS:
Device: Dexcom G6 CGM — Once discharged, the patients will be monitored by the endocrine team via routine "dashboard rounds" during working hours (8AM-5PM). Outside of dashboard rounds, management will be by exception, based on platform alarms directed to the endocrinology service.
  Other Names: Current Health Monitoring System

SUMMARY:
Patients who have experienced dysglycemia in hospital (either from diabetes, post-solid organ transplantation, medication titration, or other causes) may struggle to manage their blood glucose when discharged home. This may lead to ER visits or readmissions that could have been prevented if glucose variations were detected before reaching extremes, and the variations were contextualized with other vital sign parameters. Remote monitoring via Dexcom G6 and Current Health (vital signs) used concomitantly after discharged for the purpose of remote monitoring will be evaluated with respect to ER visits and readmissions while considering the impact and usability of the potential integrated system on the healthcare staff.

DETAILED DESCRIPTION:
This is a single-site, open label, non-randomized, pilot and feasibility study. Participants will include post-hospitalized patients who experienced inpatient dysglycemia that required management from the endocrine service (including those newly diagnosed with T1 or T2 diabetes solid organ transplantation, COPD, post respiratory infections (i.e. COVID-19), chemo patients. Approximately 40 participants will be enrolled and assigned to receive the study intervention of real time-remote monitoring (rt-RM) using the Dexcom and Current Health integrated solution.

Potential participants will be identified via the EMR by the Endocrine Team and consented prior to enrollment, 2-48 hours prior to discharge. The study team will issue them Current Health and Dexcom CGM kits and provide the necessary training. Once discharged, the patients will be monitored by the endocrine team via routine "dashboard rounds" during working hours (8AM-5PM). Outside of dashboard rounds, management will be by exception, based on platform alarms directed to the endocrinology service. Alarms will be triaged and actioned according to pre-agreed protocols, including escalation to the appropriate specialists (endocrinologist, transplant surgeon, oncologist, pneumonologist, infectious disease specialist etc.). Participants will remain enrolled in the trial until either of the two endpoints: ER visits/ readmission or 30 days post discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥21 years old
2. Treated for dysglycemia while in the acute (inpatient) period
3. With or without diabetes including patients with the following:

   * newly diagnosed T2D or T1D (LADA or other late onset)
   * post solid organ transplant
   * receiving or had received chemotherapy
   * COPD
   * Respiratory infections
4. Fit for discharge home in the opinion of the primary treating clinical team
5. Able to ambulate, or complete activities of daily living appropriate to their social care setting either on their own or with support

Exclusion Criteria:

1. Acute delirium or any other psychiatric condition that will not allow the person to participate
2. Current bleeding disorder
3. Lack of appropriate sites for CGM sensor or Current Health placement (sites must be free of large scars, skin irritation, surgical wounds, dressings, burns, anasarca, heavy tattooing etc.)
4. Any skin condition that prevents the use of CGM with adhesive
5. Known current pregnancy, breast feeding, or plan to become pregnant in the next 30 days
6. Unwilling to remove study devices prior to planned MRI and/or CT scan and reapply and wear after procedure(s) has completed.
7. Persistent atrial fibrillation
8. No access to home internet, cellular service or mobile telephone
9. Unwilling to use a study provided commercially available smartphone. The smartphones will be modified so they are only capable of hosting and running the study applications required for data collection. The modified smartphones will not be able to execute standard smartphone functionality such as internet browsing, texting, or making phone calls. Bluetooth functionality will remain intact as it is required for the approved applications to collect data.
10. Any other condition that, based on Investigator's judgment, would render the patient unsuitable to take part in the study

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Reduce amount of ER readmission in first 30 days after discharge | 30 days
  Number of participants with ER visits or readmissions as assessed by the evaluation of real time-remote monitoring (rt-RM) of blood glucose and vital signs after hospital discharge on unplanned service utilization
Pilot study satisfaction survey | 30 days or less per patient
  Questionnaire or provided summary to evaluate patient and provider satisfaction of the remote monitoring technology.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided